CLINICAL TRIAL: NCT02195492
Title: Synvisc® in With Knee Osteoarthritis: Retrospective Follow-up in Active Patients
Brief Title: Retrospective Follow-up of Synvisc® in Active Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1139.7
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — hylan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Synvisc®
  Interventions: Drug: Synvisc®

INTERVENTIONS:
Drug: Synvisc®

SUMMARY:
Retrospective collection of data, aimed at a better knowledge of the context of use of Synvisc® among the patients practising a regular activity (professional/leisure), and at evaluating the different practices and their results.

ELIGIBILITY:
Inclusion Criteria:

* use of Synvisc®
* patients practising a regular activity (professional/leisure)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: rheumatological practice
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2002-04; Primary Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Amount of medication consumed | up to 1 year
  antalgics, non-steroid anti-inflammatory drugs (NSAIDs), steroid anti-inflammatory drugs (SAIDs)

SECONDARY OUTCOMES:
Patient-assessed benefit on a 2-point verbal rating scale | up to 1 year